CLINICAL TRIAL: NCT06963580
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of MI078 Capsule in Patients With Postpartum Depression
Brief Title: Efficacy of MI078 Capsules in Treating Postpartum Depression
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing Minova Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-43
Record Dates: First submitted 2025-04-28; First posted 2025-05-09 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-04

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MI078 capsule dose 1 (Experimental): MI078 capsule dose 1
  Interventions: Drug: MI078 capsule dose 1
- MI078 capsule dose 2 (Experimental): MI078 capsule dose 2
  Interventions: Drug: MI078 capsule dose 2
- placebo (Placebo Comparator): Placebo of MI078 capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MI078 capsule dose 1 — MI078 capsule dose 1 for 3 days
  Arms: MI078 capsule dose 1
Drug: MI078 capsule dose 2 — MI078 capsule dose 2 for 3 days
  Arms: MI078 capsule dose 2
Drug: placebo — placebo for 3 days
  Arms: placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled trial. It includes three groups. Each group will enroll 24 participants. The trial aims todetermine： To evaluate the efficacy of MI078 capsules in treating postpartum depression and to explore the optimal dosing regimen for MI078 capsules.

To assess the safety of MI078 capsules in postpartum depression patients.

DETAILED DESCRIPTION:
This study employs a multicenter, randomized, double-blind, placebo-controlled parallel design. It plans to include three groups: one for the test drug at dose 1, one for the test drug at dose 2, and one for the placebo group, with 24 subjects in each group. The study consists of a screening period (D-14 to D-1), a treatment period (Day 1 to Day 4), and a follow-up period (Day 5 to Day 31). Enrolled subjects will be randomly assigned in a 1:1:1 ratio and will take the study medication for a total of 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 45 years (inclusive) with a Body Mass Index (BMI) ranging from 18.5 to 37.0 kg/m² (inclusive).
* The patient meets the diagnostic criteria for Major Depressive Disorder (MDD) as defined in the Diagnostic and Statistical Manual of Mental Disorders(DSM-5), based on the investigator's clinical evaluation. The onset of illness must occur between 28 weeks of pregnancy and 4 weeks postpartum (inclusive).
* The patient is within 9 months postpartum during the screening period.
* The total score on the HAMD17 is ≥26 during both the screening and baseline periods.
* The patient understands and voluntarily agrees to participate in the study, consents to comply with all study requirements, and is able to provide written informed consent prior to the initiation of any study-specific procedures.
* The patient is able to communicate effectively with the investigator, is willing and able to adhere to the lifestyle restrictions or requirements specified in the study protocol, and can cooperate fully in completing the trial.

Exclusion Criteria:

* Current diagnosis of another mental disorder according to DSM-5 criteria, as assessed by the investigator
* History of bipolar disorder, schizophrenia, and/or schizoaffective disorder
* History of sleep apnea
* Presence of suicidal ideation/intent, or a score >3 on Item 3 (suicide) of the HAMD17, or a response of "yes" to Item 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past 6 months, or a history of suicidal behavior within the past year
* Meeting the diagnostic criteria for treatment-resistant depression
* Continuous use of therapeutic doses of antidepressants for more than 14 days during the current episode
* Failure to discontinue psychotropic medications for at least 5 half-lives prior to the use of the study drug.
* Need for concurrent use of other psychotropic medications, such as antidepressants, antipsychotics, mood stabilizers, and sedative-hypnotics (excluding benzodiazepines), during the trial dosing period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HAM-D17 total score | up to day 31
  The Seventeen-Item Hamilton Rating Scale for Depression (HAM-D17) contains 17 individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia (initial, middle, and late), work and interests, psychomotor retardation, psychomotor agitation, anxiety (psychic and somatic), gastrointestinal symptoms, general somatic symptoms, sexual interest, hypochondriasis, insight, and weight loss. The total score ranges from 0 to 52, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
HAM-D17 response | up to day 31
  Defined as having a 50% or greater reduction from baseline in HAM-D17 total score. The total score ranges from 0 to 52, with higher scores indicating more severe depression.
HAM-D17 remission | up to day 31
  Defined as having a HAM-D17 total score ≤7. The total score ranges from 0 to 52, with higher scores indicating more severe depression
Change from baseline in the CGI-S score | up to day 31
  The CGI-S scale is a 7-point scale that requires the Investigator to assess how mentally ill is the patient at this time. 1 - normal, not at all ill; 2 - borderline mentally ill; 3 - mildly ill; 4 - moderately ill; 5 - markedly ill; 6 - severely ill; or 7 - among the most extremely ill patients
Clinical Global Impression - Improvement (CGI-I) scale positive response | up to day 31
  The CGI-I scale is a 7-point scale that requires the Investigator to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of study drug treatment. 1 - very much improved; 2 - much improved; 3 - minimally improved; 4 - no change; 5 - minimally worse; 6 - much worse; or 7 - very much worse
Change from baseline in MADRS total score | up to day 31
  The MADRS contains 10 individual items related to the following symptoms: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The total score ranges from 0 to 60, with higher scores indicating more severe depression
Change from baseline in Edinburgh Postnatal Depression Scale (EPDS) total score | up to day 31
  The Edinburgh Postnatal Depression Scale (EPDS) is a set of 10 screening questions. The total score ranges from 0 to 30, with higher scores indicating more severe depression.
Change from baseline in Hamilton Anxiety Rating Scale (HAM-A) total score | up to day 31
  The HAM-A contains 14 individual ratings related to the following symptoms: anxious mood, tension, fears, insomnia, intellectual, depressed mood, somatic (muscular), somatic (sensory), cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms, autonomic symptoms, and behavior at interview. The total score ranges from 0 to 56, with higher scores indicating more severe anxiety.
Safety Evaluation Indicators | up to day 31
  Adverse events (AEs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), clinical laboratory test, 12-lead electrocardiogram (ECG)，C-SSRS，PWC-20

CONTACTS AND LOCATIONS:
Overall Officials: huafang Li, Study Chair — Shanghai Mental Health Center
Locations (21):
- China (21):
  - The Affiliated Beijing Anding Hospital of Capital Medical University, Wuhu Hospital, Wuhu, Anhui
  - Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality
  - Xiamen Xian Yue Hospital, Xiamen, Fujian
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - The People's Hospital of Guizhou Province, Guiyang, Guizhou
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area Mental Health Center, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Affiliated Kangning Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No